CLINICAL TRIAL: NCT05012540
Title: Systemic Immune-inflammation Index (SII) And Platelet-albumin-bilirubin (PALBI) is Associated With the Prognosis of Pancreatic Cancer Surgery
Brief Title: SII And PALBI is Associated With the Prognosis of Pancreatic Cancer Surgery(SII,PALBI)
Acronym: SII
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26364
Record Dates: First submitted 2021-07-15; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; Systemic immune inflammation index; Platelet-albumin-bilirubin grade
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic inflammation and immune dysfunction play a key role in the development of tumors. The aim of the study is to investigate the predictive value of SII and PALBI grade for the patients with pancreatic cancer surgery.

DETAILED DESCRIPTION:
The systemic immune-inflammation index(SII), based on the counts of platelets, neutrophils, and lymphocytes,was first found to be related to the prognosis of patients in melanoma12, and was subsequently confirmed in malignant tumors such as hepatocellular carcinoma13,and lung cancer12. A retrospective multicenter cohort study showed that bilirubin levels can interfere some inflammation index'prognosis of PDAC7.The platelet-albumin-bilirubin (platelet-albumin-bilirubin, PALBI) grade as a prognostic indicator of inflammation has been found in recent years, and its role has been confirmed in patients with liver cirrhosis14,15 and hepatocellular carcinoma 16, but there is no research to verify its role in patients with pancreatic cancer. This study aims to verify the predictive value of systemic immune inflammation index (SII) and platelet-albumin-bilirubin grade (PALBI) for the prognosis of patients with pancreatic cancer surgery, and to explore the significance of other inflammatory indicators in the overall survival(OS) and disease-free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old; It was diagnosed as pancreatic cancer by clinical manifestations, laboratory examination indexes, and pathology, and then surgically removed; Agree to participate in this study and sign an informed consent form;

Exclusion Criteria:

All kinds of acute or chronic inflammation, infectious diseases and blood system diseases; Metastasis of tumors in other parts; Benign pancreatic diseases such as chronic pancreatitis and autoimmune pancreatitis; Periampullary tumors without pancreatic cancer; Suspicious pancreatic cancer patients who cannot be diagnosed; Refuse to follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age≥18 years old
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The overall survival | 2013.8-2019.12
  The overall survival（OS）was defined as time between primary surgery and the patients' death. Death from other cause than PDAC or survival until the end of the observation period was considered as censored observations